CLINICAL TRIAL: NCT02647749
Title: Non-invasive Mapping of Rhythm Disorders
Acronym: CARRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2015/01
Record Dates: First submitted 2015-11-05; First posted 2016-01-06 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Rhythm Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 : Cardiac rythm radiofrequency ablation (Experimental): Prospective recruitment
  Interventions: Device: Cardioinsight® mapping system
- Group 1: Implantation or programming of a pacemaker (Experimental): Prospective recruitment
  Interventions: Device: Cardioinsight® mapping system
- Group 1: Risk of serious arrhythmias or sudden death (Experimental): Prospective recruitment
  Interventions: Device: Cardioinsight® mapping system
- Group 2: Cardiac rythm radiofrequency ablation (Active Comparator): Retrospective recruitment
  Interventions: Other: Conventional method without non-invasive mapping
- Group 2 : Implantation or programming of a pacemaker (Active Comparator): Retrospective recruitment
  Interventions: Other: Conventional method without non-invasive mapping
- Group 2 : Risk of serious arrhythmias or sudden death (Active Comparator): Retrospective recruitment
  Interventions: Other: Conventional method without non-invasive mapping

INTERVENTIONS:
Device: Cardioinsight® mapping system
  Arms: Group 1 : Cardiac rythm radiofrequency ablation; Group 1: Implantation or programming of a pacemaker; Group 1: Risk of serious arrhythmias or sudden death
Other: Conventional method without non-invasive mapping
  Arms: Group 2 : Implantation or programming of a pacemaker; Group 2 : Risk of serious arrhythmias or sudden death; Group 2: Cardiac rythm radiofrequency ablation

SUMMARY:
This current care protocol follows the biomedical research protocol entitled "Non-invasive mapping of the heart ECG high amplification" that demonstrated the clinical value of noninvasive Cardioinsight® mapping system.

Guide the management of patients hospitalized for cardiac rhythm radiofrequency ablation of cardiac arrhythmias, implantation or programming of a pacemaker, or assess the risk of serious arrhythmias or sudden death, with the currently used non-invasive mapping routine. The results obtained with non-invasive mapping will be compared with those obtained with the conventional method without non-invasive mapping.

DETAILED DESCRIPTION:
This current care protocol is for 3 groups of patients :

1. Role of mapping arrhythmias before radiofrequency ablation :

   Radiofrequency ablation is a treatment of atrial or ventricular arrhythmias resistant to drug treatment. The electrocardiogram does not allow a full diagnosis of arrhythmias and it appears difficult to get a comprehensive and simultaneous view of cardiac activity during invasive maps. The Investigators have demonstrated the feasibility of mapping atrial fibrillation and its usefulness to guide radiofrequency ablation. The non-invasive mapping would allow a better understanding of complex cardiac arrhythmias mechanism (atrial fibrillation, ventricular tachycardia and ventricular fibrillation in particular), would identify the arrhythmogenic sites and thus facilitate radiofrequency ablation.
2. Optimizing the site of implantation of cardiac pacing leads and programming the pacemaker:

   The optimal position of the cardiac pacing leads may vary from one patient to another and the current choice of implantation sites is essentially guided by imaging and does not use power requirements because of the inadequacies of the ECG standard. The Investigators have already demonstrated the usefulness of non-invasive mapping in the selection of potential responders to cardiac resynchronization therapy. The non-invasive mapping would study the cardiac electrical activation in order to determine the optimal pacing sites and optimum programming according to each patient and thus improve the clinical response to pacing.
3. Role diagnostic and prognostic for patients referred for evaluation of the risk of occurrence of a serious rhythm disorder or sudden death :

The possibility to identify electrically abnormal areas either during the activation, or during cardiac repolarization with the high-resolution ECG is an indication of myocardial pathology that can be both unapparent on standard ECG and inaccessible to imaging techniques (ultrasound, CT or MRI). It is likely that such electrical anomalies are early diagnostic features of heart disease that will later be apparent. Such anomalies can also have an adverse prognostic weight (risk of arrhythmias or sudden death) that can be corrected if it is highlighted. Non-invasive mapping seems particularly important in patients with unexplained symptoms by conventional tests (palpitations or discomfort - syncope). It will also be applicable to patients with heart disease (myocardial infarction, cardiomyopathy) in search of localized electrical disorders that can be an originating site of arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Oral agreement of the patient or of the holder of parental responsibility after reading the informed consent form.
* Patients with the following 3 conditions :
* Ablation of drugs rebels arrhythmias.
* Or implantation or programming of a pacemaker (pacemaker or defibrillator)
* Or symptoms and / or cardiopathy with risk of sudden death.

Exclusion Criteria:

* Pregnancy and lactation.
* Patients unable to give oral agreement.
* Inconsistent patient's morphology with the establishment of the electrode jacket

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Arrhythmia termination during ablation guided by the Cardioinsight® mapping system | Day 1
Variation of dP/dT measurement between baseline and after implantation or programmation of a pacemaker guided by the Cardioinsight® mapping system | Day 1
  In mmHg/s
Measurement of the activation-recovery interval defined as the interval between a local depolarization time and repolarization time for patients referred for evaluation of the risk of occurrence of a serious rhythm disorder or sudden death | Day 1
  In ms

SECONDARY OUTCOMES:
Arrhythmia recurrence at 1 year after ablation guided by the Cardioinsight® mapping system | Year 1
For patients referred for implantation or programming of a pacemaker: Comparison of 6 Minutes Walk Test performed before and 6 months after implantation and/or programmation guided by the Cardioinsight® mapping system | Month 6
  In meters
For patients referred for implantation or programming of a pacemaker: Comparison of left ventricular ejection fraction performed before and 6 months after implantation and/or programmation guided by the Cardioinsight® mapping system | Month 6
  In percentage
Occurence of syncope, aborted sudden death or sudden death during follow-up for patients referred for evaluation of the risk of occurrence of a serious rhythm disorder or sudden death | Year 1, year 4 at most

CONTACTS AND LOCATIONS:
Overall Officials: Michel HAÏSSAGUERRE, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France